CLINICAL TRIAL: NCT06731881
Title: Leveraging Photodynamic Therapy to Inhibit Microorganisms - Assessing the Efficacy of Photodynamic Therapy for Preventing Surgical Site Infections in Nasal Surgery Patients: A Pilot Study
Brief Title: Assessing the Efficacy of Photodynamic Therapy for Preventing Surgical Site Infections
Acronym: LIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRAS345142
Record Dates: First submitted 2024-12-11; First posted 2024-12-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Surgery; Nasal Disease; Light; Therapy, Complications
Keywords: nasal surgery; nasal photodisinfection; decolonisation; surgical site infection
MeSH Terms: conditions — Nose Diseases; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: A randomised, interventional proof of concept pilot trial in which patients undergoing nasal surgery will be selected for either photodisinfection therapy with the Steriwave™ ND System, or control with nares swabbed with 'photosensitizer formulation' (0.01% methylene blue with 0.25% chlorhexidine solution) prior to surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodisinfection (Active Comparator): The photodisinfection product consists of a CE-marked light source (SW4000), a disposable single-use nasal light diffuser, and a single-use photosensitiser applicator that can be used in hospital settings.
  Interventions: Device: Nasal PDT; Other: Standard follow-up; Diagnostic Test: Nasal culture; Diagnostic Test: Flexible nasendoscopy; Other: In-person review; Other: Telephone Follow-up
- Control (Active Comparator): The control group will have nares swabbed with 'photosensitizer formulation' (0.01% methylene blue with 0.25% chlorhexidine solution) prior to surgery.
  Interventions: Combination Product: Photosensitizer formulation only; Other: Standard follow-up; Diagnostic Test: Nasal culture; Diagnostic Test: Flexible nasendoscopy; Other: In-person review; Other: Telephone Follow-up

INTERVENTIONS:
Device: Nasal PDT — Two two-minute cycles will be provided by a member of the research team in the pre-operative area on the day of surgery. A saturated swab containing 0.01% methylene blue and 0.25% chlorhexidine gluconate will be applied to nares, which is then activated by light.
  Other Names: Steriwave (SW4000)
  Arms: Photodisinfection
Combination Product: Photosensitizer formulation only — Nares will be swabbed with Photosensitizer formulation (0.01% methylene blue with 0.25% chlorhexidine solution). Nasal swab cultures will be obtained before control swabbing and converted to colony-forming units to measure bacterial burden at baseline, and after treatment (2 weeks +/- 7 days). Sinonasal mucosal inflammation using the Flexible Nasendoscopy Endoscopic LK Score will also be obtained before treatment at 2 weeks (+/-7 days).
  Arms: Control
Other: Standard follow-up — All patients will receive standard post-operative wound follow up. This might include being advised to contact the GP or the hospital if there are any wound problems and, or, being invited to an out-patient clinic appointment.
Diagnostic Test: Nasal culture — Nasal swab cultures will be obtained before Nasal PDT or control swabbing and converted to colony-forming units to measure bacterial burden at baseline, and after treatment (2 weeks +/- 7 days).
Diagnostic Test: Flexible nasendoscopy — Sinonasal mucosal inflammation using the Flexible Nasendoscopy Endoscopic Lund-Kennedy (LK) Score will also be obtained before Nasal PDT or control swabbing and at 2 weeks (+/-7 days).
Other: In-person review — On Week 2 (±7 days), the participant will undergo an in-person review conducted in the ENT Outpatient department, 2nd floor Southwark wing, Guy's Hospital by the CI, PI or Co-investigator. During this appointment, concomitant medications and use of post-operative antibiotics will be reviewed.
Other: Telephone Follow-up — On day 30, the research nurse will telephone participants from the ENT research office.
  * Review of adverse events/adverse device effects
  * Review of concomitant medications
  * Signs and symptoms post-surgery
  * Nasal washout
  * Record any use of post-operative antibiotics, both local and systemic

SUMMARY:
This is a randomised, unblinded interventional device proof of concept pilot trial in which patients undergoing nasal surgery will be selected for either photodisinfection therapy (PDT) with the Steriwave™ ND System, or control with nares swabbed with 'photosensitizer formulation' preoperatively.

This trial will primarily assess the safety and efficacy of nasal photodisinfection treatment in decreasing post-operative events in patients undergoing nasal surgery. After signing informed consent, and before surgery, participants will receive a baseline culture of the anterior nares to determine nasal bacterial colonization and will have a flexible nasendoscopy to determine their Lund-Kennedy (LK) endoscopic score. Subjects will then be randomised to nasal PDT (which includes two applications of 'photosensitizer formulation' [0.01% methylene blue with 0.25% chlorhexidine solution], two minutes apart), along with light therapy, or control with nares swabbed twice with 'photosensitizer formulation' with two minutes in between (no light therapy). Following treatment, participants will be re-cultured (2 weeks after the surgery ± 7 days) and reviewed for antibiotic use and surgical site infection (SSI) using LK endoscopic scoring. At 30 days, all participants will be followed up by telephone to review if they received antibiotics for presumed postoperative infection. Standard post-operative care will be provided according to the type of surgery performed. Any required interventions post-operatively will be documented.

DETAILED DESCRIPTION:
Preoperative nasal decolonisation has been shown to achieve significant reductions in surgical site infections at sites remote from the nasal cavity. It would therefore seem to have great potential in reducing the risk of post-operative infections after sinonasal surgery, and therefore reduce antibiotic usage. If surgeons have confidence in the treatment, those that routinely prescribe prophylactic antibiotics may also be pursued to change their practice.

The aim of this study is to assess the efficacy and safety of photodisinfection therapy versus control with nares swabbed with 'photosensitizer formulation' (0.01% methylene blue with 0.25% chlorhexidine solution) to reduce the antibiotics usage for presumed SSI inpatients undergoing nasal surgery. The investigators hypothesise that preoperative photodisinfection will demonstrate greater efficacy compared to control with nares swabbed with 'photosensitizer formulation' (0.01% methylene blue with 0.25% chlorhexidine solution) in reducing the usage of antibiotics for presumed surgical site infection (SSI) among patients undergoing nasal surgery.

The investigators will also further evaluate the effectiveness of nasal decolonisation in eliminating colonization of the anterior nares with S. aureus and other potentially pathogenic microbes. The anterior nares are often considered the primary reservoir of S. aureus and other pathogens on the body (36). Therefore, this product could play an important role in helping to eliminate the anterior nares as a pathogen reservoir in surgical patients.

This study is meant to provide further safety, efficacy, and methodological data, but is not intended to establish definitive statistical significance. If required, this study will support a subsequent larger study that would establish statistical significance for the reduction of surgical site infections, but which is currently not the subject of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years
* Patients scheduled to undergo elective:

  * Endoscopic Sinus Surgery (ESS) with or without adjunctive Septoplasty and/or Turbinoplasty
  * Septoplasty with or without adjunctive Turbinoplasty
  * Closed Septoplasty with or without adjunctive Turbinoplasty
* Judged by the Investigator as suitable for participation in the study without safety concerns based on medical history and physical examination
* Willing and able to provide written informed consent prior to participation in the clinical investigation
* Willing and able to comply with all study related procedures

Exclusion Criteria:

-• Patients undergoing open septorhinoplasty, anterior or septal biopsies, or post cautery

* Congenital or acquired immunodeficiency, bone marrow disease, diabetes, autoimmune conditions requiring immunosuppressive treatment, any immunosuppressive medication at the time of consent or within the last 4 weeks before randomisation
* Primary or secondary ciliary dyskinesia, cystic fibrosis
* Patients who have received antibiotics within a week before randomisation
* Patients who receive prophylactic antibiotics or antibiotics prior to discharge
* Systemic steroid treatment less than 4 weeks before randomisation
* History of frequent nose bleeds, or a condition that increases the risk of excessive bleeding
* Undergoing active cancer treatment at time of consent/ or planning to start cancer treatment within trial period or completed cancer treatment within the last 4 weeks
* Any disease, condition (medical or surgical), or drug or alcohol abuse, which, in the opinion of the investigator, might compromise the study results, or would place the patient at increased risk of infection
* Previously treated with radiation on the face, head, or neck regions
* Female patients who are pregnant or breastfeeding at the time of consent
* Received a study drug in a clinical trial for an investigational drug within the previous 30 days from consent, or 5 half-lives, whichever is longer
* Used antimicrobial wash or wipes within 7 days of randomisation or during the study period
* Patients with allergies / hypersensitivity to methylene blue, polymethyl methacrylate (PMMA), or to chlorhexidine gluconate (CHG)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Antibiotic usage in number and percentages | 30 days
  The proportion of patients requiring antibiotic therapy for presumed surgical site infections (SSIs) within 30 days after undergoing nasal surgery. Specifically, the intention is to compare those who received preoperative PDT with those in the control group.

SECONDARY OUTCOMES:
Incidence of surgical site infection | 30 days
  The proportion of patients developing a postoperative infection within 30 days of surgery, defined by the presence of sinus purulence (Lund-Kennedy score of 2: 'Thick and purulent discharge') on nasal endoscopy and requiring antibiotic treatment.
Lund-Kennedy Score Assessment | 30 days
  The change in Lund-Kenned (LK) scores from baseline during the study period, as measured by flexible nasendoscopy, in patients who received preoperative PDT compared to those in the control group.
  Each side is graded on an ordinal scale from 0-2, with higher scores indicating worse disease.
Bacterial Nasal Culture Rates | 30 days
  The percentage of patients with positive bacterial cultures (S. aureus and Group A Streptococcus) from nasal swabs during the study period, comparing the PDT group with the control group.

OTHER OUTCOMES:
Safety of PDT | 30 days
  The incidence of adverse events or complications (e.g., nasal irritation, bleeding, discomfort) associated with the nasal photodisinfection procedure, as reported by patients and assessed by clinical examination during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Hopkins, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The trial will be conducted in accordance with the Data Protection Act 2018. The chief investigator will ensure that participant's anonymity is maintained throughout the study and following completion of the study.
  Pseudonymised data will be shared with the study Statistician who is an employee of the Trust and member of the study team. It will be extracted from REDCap and sent via encrypted email in a locked Excel document. After the analysis the data will be archived in Iron Mountain.
  No data will be shared outside of GSTT during the course of the study.
  Data will not be shared with the device manufacturer.

REFERENCES:
- [Background] Psaltis AJ, Li G, Vaezeafshar R, Cho KS, Hwang PH. Modification of the Lund-Kennedy endoscopic scoring system improves its reliability and correlation with patient-reported outcome measures. Laryngoscope. 2014 Oct;124(10):2216-23. doi: 10.1002/lary.24654. Epub 2014 Apr 2. PMID 24615873
- [Background] Carrie S, O'Hara J, Fouweather T, Homer T, Rousseau N, Rooshenas L, Bray A, Stocken DD, Ternent L, Rennie K, Clark E, Waugh N, Steel AJ, Dooley J, Drinnan M, Hamilton D, Lloyd K, Oluboyede Y, Wilson C, Gardiner Q, Kara N, Khwaja S, Leong SC, Maini S, Morrison J, Nix P, Wilson JA, Teare MD. Clinical effectiveness of septoplasty versus medical management for nasal airways obstruction: multicentre, open label, randomised controlled trial. BMJ. 2023 Oct 18;383:e075445. doi: 10.1136/bmj-2023-075445. PMID 37852641
- [Background] Rochon M, Jawarchan A, Ingusan S, Cariaga K and Morais C. 'Project ID007672: Clinical audit of patient-reported antibiotics for wound problems following surgery and review of alternative strategies'. 2023 Feb 25. Unpublished.
- [Background] Street CN, Pedigo L, Gibbs A, Loebel NG. Antimicrobial photodynamic therapy for the decolonization of methicillin-resistant Staphylococcus aureus from the anterior nares, Proc. SPIE 7380, Photodynamic Therapy: Back to the Future, 73803B (13 July 2009); https://doi.org/10.1117/12.828279
- [Background] Ontario Health (Quality). Pre-surgical Nasal Decolonization of Staphylococcus aureus: A Health Technology Assessment. Ont Health Technol Assess Ser. 2022 Aug 23;22(4):1-165. eCollection 2022. PMID 36160757
- [Background] Hsiao CJ, Paulson JN, Singh S, Mongodin EF, Carroll KC, Fraser CM, Rock P, Faraday N. Nasal Microbiota and Infectious Complications After Elective Surgical Procedures. JAMA Netw Open. 2021 Apr 1;4(4):e218386. doi: 10.1001/jamanetworkopen.2021.8386. PMID 33914049
- [Background] Bryce E, Wong T, Forrester L, Masri B, Jeske D, Barr K, Errico S, Roscoe D. Nasal photodisinfection and chlorhexidine wipes decrease surgical site infections: a historical control study and propensity analysis. J Hosp Infect. 2014 Oct;88(2):89-95. doi: 10.1016/j.jhin.2014.06.017. Epub 2014 Aug 1. PMID 25171975
- [Background] Braham P, Herron C, Street C, Darveau R. Antimicrobial photodynamic therapy may promote periodontal healing through multiple mechanisms. J Periodontol. 2009 Nov;80(11):1790-8. doi: 10.1902/jop.2009.090214. PMID 19905948
- [Background] Andersen R, Loebel N, Hammond D, Wilson M. Treatment of periodontal disease by photodisinfection compared to scaling and root planing. J Clin Dent. 2007;18(2):34-8. PMID 17508621
- [Background] Andersen R, Loebel N. Photodynamic Disinfection in the Treatment of Chronic Adult Periodontitis: A Multicentre Clinical Trial. J Dent Health Oral Disord Ther 2017, 8(4): 00289. DOI: 10.15406/jdhodt.2017.08.00289
- [Background] Dinis-Ribeiro M, Moreira-Dias L. There is no clinical evidence of consequences after methylene blue chromoendoscopy. Gastrointest Endosc. 2008 Jun;67(7):1209. doi: 10.1016/j.gie.2007.12.043. No abstract available. PMID 18513562
- [Background] ASGE Technology Committee; Thosani N, Abu Dayyeh BK, Sharma P, Aslanian HR, Enestvedt BK, Komanduri S, Manfredi M, Navaneethan U, Maple JT, Pannala R, Parsi MA, Smith ZL, Sullivan SA, Banerjee S. ASGE Technology Committee systematic review and meta-analysis assessing the ASGE Preservation and Incorporation of Valuable Endoscopic Innovations thresholds for adopting real-time imaging-assisted endoscopic targeted biopsy during endoscopic surveillance of Barrett's esophagus. Gastrointest Endosc. 2016 Apr;83(4):684-98.e7. doi: 10.1016/j.gie.2016.01.007. Epub 2016 Feb 11. PMID 26874597
- [Background] Millson CE, Thurrell W, Buonaccorsi G, et al. The effect of low power laser light at different doses on gastric mucosa sensitised with methylene blue, hematoporphyrin derivative or toluidine blue. Laser Med Sci 1997; 12:145-150.
- [Background] Sturmey RG, Wild CP, Hardie LJ. Removal of red light minimizes methylene blue-stimulated DNA damage in oesophageal cells: implications for chromoendoscopy. Mutagenesis. 2009 May;24(3):253-8. doi: 10.1093/mutage/gep004. Epub 2009 Feb 13. PMID 19218330
- [Background] Olliver JR, Wild CP, Sahay P, Dexter S, Hardie LJ. Chromoendoscopy with methylene blue and associated DNA damage in Barrett's oesophagus. Lancet. 2003 Aug 2;362(9381):373-4. doi: 10.1016/s0140-6736(03)14026-3. PMID 12907012
- [Background] Davies J, Burke D, Olliver JR, Hardie LJ, Wild CP, Routledge MN. Methylene blue but not indigo carmine causes DNA damage to colonocytes in vitro and in vivo at concentrations used in clinical chromoendoscopy. Gut. 2007 Jan;56(1):155-6. doi: 10.1136/gut.2006.107300. No abstract available. PMID 17172595
- [Background] Canto MI, Setrakian S, Petras RE, Blades E, Chak A, Sivak MV Jr. Methylene blue selectively stains intestinal metaplasia in Barrett's esophagus. Gastrointest Endosc. 1996 Jul;44(1):1-7. doi: 10.1016/s0016-5107(96)70221-3. PMID 8836709
- [Background] Kohli Y, Pfeiffer CJ, Kutty KP, Barrowman JA, Heughan C, Kepkay DL. Endoscopic diagnosis of intestinal metaplasia in Canada and Japan. J Clin Gastroenterol. 1981;3 Suppl 1:29-33. doi: 10.1097/00004836-198100031-00006. PMID 7328294
- [Background] Suzuki S, Suzuki H, Endo M, Takemoto T, Kondo T. Endoscopic diagnosis of early cancer and intestinal metaplasia of the stomach by dyeing. Int Surg. 1973 Sep;58(9):639-42. No abstract available. PMID 4744424
- [Background] Shah-Khan MG, Lovely J, Degnim AC. Safety of methylene blue dye for lymphatic mapping in patients taking selective serotonin reuptake inhibitors. Am J Surg. 2012 Nov;204(5):798-9. doi: 10.1016/j.amjsurg.2012.02.004. Epub 2012 May 9. PMID 22575397
- [Background] FDA Drug Safety Communication dated 26 July 2011 - accessed on 31 January 2019 at - http://www.fda.gov/Drugs/DrugSafety/ucm263190.htm
- [Background] Dewachter P, Mouton-Faivre C, Trechot P, Lleu JC, Mertes PM. Severe anaphylactic shock with methylene blue instillation. Anesth Analg. 2005 Jul;101(1):149-50, table of contents. doi: 10.1213/01.ANE.0000153497.60047.80. PMID 15976222
- [Background] Bezu C, Coutant C, Salengro A, Darai E, Rouzier R, Uzan S. Anaphylactic response to blue dye during sentinel lymph node biopsy. Surg Oncol. 2011 Mar;20(1):e55-9. doi: 10.1016/j.suronc.2010.10.002. Epub 2010 Nov 11. PMID 21074413
- [Background] Masannat YA, Hanby A, Horgan K, Hardie LJ. DNA damaging effects of the dyes used in sentinel node biopsy: possible implications for clinical practice. J Surg Res. 2009 Jun 15;154(2):234-8. doi: 10.1016/j.jss.2008.07.039. Epub 2008 Sep 4. PMID 19181339
- [Background] Wainwright M, Crossley KB. Methylene Blue--a therapeutic dye for all seasons? J Chemother. 2002 Oct;14(5):431-43. doi: 10.1179/joc.2002.14.5.431. PMID 12462423
- [Background] Silva ZS Jr, Bussadori SK, Fernandes KP, Huang YY, Hamblin MR. Animal models for photodynamic therapy (PDT). Biosci Rep. 2015 Sep 28;35(6):e00265. doi: 10.1042/BSR20150188. PMID 26415497
- [Background] Dai T, Tegos GP, Zhiyentayev T, Mylonakis E, Hamblin MR. Photodynamic therapy for methicillin-resistant Staphylococcus aureus infection in a mouse skin abrasion model. Lasers Surg Med. 2010 Jan;42(1):38-44. doi: 10.1002/lsm.20887. PMID 20077489
- [Background] Zolfaghari PS, Packer S, Singer M, Nair SP, Bennett J, Street C, Wilson M. In vivo killing of Staphylococcus aureus using a light-activated antimicrobial agent. BMC Microbiol. 2009 Feb 4;9:27. doi: 10.1186/1471-2180-9-27. PMID 19193212
- [Background] Fang CH, Fastenberg JH, Fried MP, Jerschow E, Akbar NA, Abuzeid WM. Antibiotic use patterns in endoscopic sinus surgery: a survey of the American Rhinologic Society membership. Int Forum Allergy Rhinol. 2018 Apr;8(4):522-529. doi: 10.1002/alr.22085. Epub 2018 Jan 15. PMID 29334432
- [Background] Abuzeid W, Shah S, Hawn V, Fang C, Akbar N. Postoperative infection rates and associated factors following endoscopic sinus surgery. Int Forum Allergy Rhinol 2019; 9(10);1227. First Published online: August 20, 2019
- [Background] Virkkula P, Makitie AA, Vento SI. Surgical outcome and complications of nasal septal perforation repair with temporal fascia and periosteal grafts. Clin Med Insights Ear Nose Throat. 2015 Apr 29;8:7-11. doi: 10.4137/CMENT.S23230. eCollection 2015. PMID 25987852
- [Background] Dabrowska-Bien J, Skarzynski PH, Gwizdalska I, Lazecka K, Skarzynski H. Complications in septoplasty based on a large group of 5639 patients. Eur Arch Otorhinolaryngol. 2018 Jul;275(7):1789-1794. doi: 10.1007/s00405-018-4990-8. Epub 2018 May 16. PMID 29770875
- [Background] von Eiff C, Becker K, Machka K, Stammer H, Peters G. Nasal carriage as a source of Staphylococcus aureus bacteremia. Study Group. N Engl J Med. 2001 Jan 4;344(1):11-6. doi: 10.1056/NEJM200101043440102. PMID 11136954
- [Background] Kuehnert MJ, Kruszon-Moran D, Hill HA, McQuillan G, McAllister SK, Fosheim G, McDougal LK, Chaitram J, Jensen B, Fridkin SK, Killgore G, Tenover FC. Prevalence of Staphylococcus aureus nasal colonization in the United States, 2001-2002. J Infect Dis. 2006 Jan 15;193(2):172-9. doi: 10.1086/499632. Epub 2005 Dec 15. PMID 16362880
- [Background] Khorvash F, Abdi F, Kashani HH, Naeini FF, Narimani T. Staphylococcus aureus in Acne Pathogenesis: A Case-Control Study. N Am J Med Sci. 2012 Nov;4(11):573-6. doi: 10.4103/1947-2714.103317. PMID 23181229
- [Background] Zanger P, Nurjadi D, Vath B, Kremsner PG. Persistent nasal carriage of Staphylococcus aureus is associated with deficient induction of human beta-defensin 3 after sterile wounding of healthy skin in vivo. Infect Immun. 2011 Jul;79(7):2658-62. doi: 10.1128/IAI.00101-11. Epub 2011 Apr 4. PMID 21464083
- [Background] Wertheim HF, Melles DC, Vos MC, van Leeuwen W, van Belkum A, Verbrugh HA, Nouwen JL. The role of nasal carriage in Staphylococcus aureus infections. Lancet Infect Dis. 2005 Dec;5(12):751-62. doi: 10.1016/S1473-3099(05)70295-4. PMID 16310147
- [Background] National Healthcare Safety Network, Centers for Disease Control and Prevention. Surgical site infection (SSI) event. http://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf. Published January 2017.
- [Background] Bachert C, Pawankar R, Zhang L, Bunnag C, Fokkens WJ, Hamilos DL, Jirapongsananuruk O, Kern R, Meltzer EO, Mullol J, Naclerio R, Pilan R, Rhee CS, Suzaki H, Voegels R, Blaiss M. ICON: chronic rhinosinusitis. World Allergy Organ J. 2014 Oct 27;7(1):25. doi: 10.1186/1939-4551-7-25. eCollection 2014. PMID 25379119
- [Background] Annys E, Jorissen M. Short term effects of antibiotics (Zinnat) after endoscopic sinus surgery. Acta Otorhinolaryngol Belg. 2000;54(1):23-8. PMID 10719590
- [Background] Fernandes SV. Postoperative care in functional endoscopic sinus surgery? Laryngoscope. 1999 Jun;109(6):945-8. doi: 10.1097/00005537-199906000-00020. PMID 10369288
- [Background] Jorissen M, Bachert C. Effect of corticosteroids on wound healing after endoscopic sinus surgery. Rhinology. 2009 Sep;47(3):280-6. doi: 10.4193/Rhin08.227. PMID 19839251